CLINICAL TRIAL: NCT02333773
Title: Irreversible Electroporation(IRE) For Unresectable Portal Venous Tumor Emboli: Phase I and Phase II Clinical Trial
Brief Title: Irreversible Electroporation(IRE) For Unresectable Portal Venous Tumor Emboli
Acronym: IRE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fuda Cancer Hospital, Guangzhou (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ZhangZhikai-IRE-01
Record Dates: First submitted 2015-01-06; First posted 2015-01-07 (Estimated); Last update posted 2021-09-05 (Actual); Status verified 2019-05

CONDITIONS: Liver Cancer
Keywords: irreversible electroporation; Portal venous tumor emboli
MeSH Terms: conditions — Liver Neoplasms | interventions — Electroporation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group A (Experimental): irreversible electroporation with voltage in level A for Unresectable Portal Venous Tumor Emboli
  Interventions: Procedure: Irreversible electroporation (IRE)
- Group B (Experimental): irreversible electroporation with voltage in level B for Unresectable Portal Venous Tumor Emboli
  Interventions: Procedure: Irreversible electroporation (IRE)
- Group C (Experimental): irreversible electroporation with voltage in level C for Unresectable Portal Venous Tumor Emboli
  Interventions: Procedure: Irreversible electroporation (IRE)

INTERVENTIONS:
Procedure: Irreversible electroporation (IRE) — Irreversible Electroportion For Unresectable Portal venous tumor emboli guide with ultrasound or/and CT.
  Other Names: NanoKnife

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of irreversible electroporation (IRE) for unresectable Portal venous tumor emboli.

DETAILED DESCRIPTION:
By enrolling patients with unresectable Portal venous tumor emboli adapted to enrolled criteria, this study will document for the first time the safety and the short and long term efficacy of percutaneous or intraoperative IRE for unresectable Portal venous tumor emboli.

ELIGIBILITY:
Inclusion Criteria:

* Liver cancer diagnosed by positive biopsy or non-invasive criteria,
* Liver cancer with Portal venous tumor emboli,
* Not suitable for surgical resection or transplantation,
* Child-Pugh class A,B
* Eastern Cooperative Oncology Group (ECOG) score of 0-1,
* A prothrombin time ratio > 50%,
* Platelet count > 80x10^9/L,
* Ability of patient to stop anticoagulant and anti-platelet therapy for seven days prior to and seven days post NanoKnife procedure,
* Able to comprehend and willing to sign the written informed consent form (ICF),
* Have a life expectancy of at least 3 months.

Exclusion Criteria:

* Cardiac insufficiency, ongoing coronary artery disease or arrhythmia,
* Any active implanted device (eg Pacemaker),
* Women who are pregnant or women of child-bearing potential who are not using an acceptable method of contraception,
* Have received treatment with an investigational agent/ procedure within 30 days prior to treatment with the NanoKnife™ LEDC System,
* Are in the opinion of the Investigator unable to comply with the visit schedule and protocol evaluations.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Safety (adverse effects) | 6 month
  adverse effects

SECONDARY OUTCOMES:
Efficacy (percentage of lesions that show no sign of recurrence 12 months after IRE) | 12 months
  The primary objective of this project is to evaluate the efficacy (percentage of lesions that show no sign of recurrence 12 months after IRE）
Voltage (A minimum and maximum range of voltage for safe and effective IRE) | 3 months
  A minimum and maximum range of voltage for safe and effective IRE will be analyzed for optimal choice.
Progress free disease (PFS) | 12 months
  Patients will be followed for 12 months after IRE for PFS assessing.
Overall survival (OS) | 36 months
  Patients will be followed for 36 months after IRE for OS analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Lizhi Niu, PHD, Study Chair — Fuda Cancer Hospital
Locations (1):
- Fuda Cancer Hospital, Guangzhou, Guangdong, China